CLINICAL TRIAL: NCT01768130
Title: Variability in Thermal Thresholds in Patients With Persistent Pain After Open Inguinal Herniotomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Joakim Bischoff, MD, Rigshospitalet, Denmark
Other Study IDs: H-2-2011-023
Record Dates: First submitted 2013-01-07; First posted 2013-01-15 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Persistent Pain After Open Inguinal Herniotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will investigate the test-retest variability of thermal thresholds in patients with persistent pain after open inguinal herniotomy. Sensory mapping with a cool metal roller delineated an area with cool sensory dysfunction on the painful site. In this area and in a contralateral area as a control, 5 sites were outlined, including the point of maximum pain. In these total 10 sites warmth detection threshold (WDT), cool detection threshold (CDT) and heat pain threshold (HPT) were assessed using quantitative sensory testing. Tests were repeated after a 4-6 weeks interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent pain after open inguinal herniotomy
* Age > 18 years

Exclusion Criteria:

* Cognitive impairment
* Drug or alcohol abuse
* Bilateral inguinal hernia operation
* Nerve injury from other causes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with persistent pain after open inguinal herniotomy
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Test- retest variability of thermal thresholds. | At baseline and retest 4-6 weeks later
  Analysis of agreement (Bland-Altman) and reliability (intraclass correlation coefficients) of thermal threshold test- retest data assessed at baseline and after 4-6 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Ø, Denmark